CLINICAL TRIAL: NCT03500146
Title: Sexual Function Trial of Overactive Bladder: Medication Versus PTNS
Acronym: STOMP
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Indiana University (Other); University of Oklahoma (Other); University of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-248
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Female Sexual Dysfunction; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Cholinergic Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal sexual function: Patients with an overall FSFI score equal to or above 26.5 will be in the normal sexual function group. Patients in both groups will be treated with an overactive bladder treatment, either anticholinergics, beta-agonists or PTNS.
  Interventions: Drug: Anticholinergic; Procedure: PTNS
- Low sexual function: Female sexual dysfunction is defined as an overall FSFI score below 26.5, patients meeting this criteria will be in the low sexual function group. Patients in both groups will be treated with an overactive bladder treatment, either anticholinergics, beta-agonists or PTNS.
  Interventions: Drug: Anticholinergic; Procedure: PTNS

INTERVENTIONS:
Drug: Anticholinergic — Patients prescribed medication for OAB
  Other Names: Beta-agonists
Procedure: PTNS — Patients prescribed PTNS for OAB

SUMMARY:
Sexual dysfunction affects approximately 45% of women with an even greater incidence reported in women with overactive bladder symptoms, despite this there is a lack of FDA approved treatments for sexual dysfunction in this population. While both medical therapy and electrical neuromodulation have been shown to improve urinary function as well as sexual function, there is a dearth of literature about their comparative effectiveness in the latter. The purpose of this study is to examine the comparative effectiveness of neuromodulation via percutaneous tibial nerve stimulation (PTNS) and medical therapy with anticholinergics or beta-agonists in improving female sexual function. This will be a prospective multi-center cohort study comparing improvement in sexual function as measured by the female sexual function index (FSFI). It is hypothesized that PTNS will improve sexual function to a greater degree than medical therapy as there may be mechanisms by which PTNS directly affects sexual function. Enhanced understanding of the effects of neuromodulation and medical therapy on sexual function may allow for improved patient selection and better outcomes which may lead to widespread use of neuromodulation for female sexual dysfunction.

DETAILED DESCRIPTION:
Specific aims:

Primary aim:

Aim 1: To determine if there is greater improvement in female sexual function as measured by the female sexual function index (FSFI) with percutaneous tibial nerve stimulation (PTNS) as compared to medical therapy (MT).

Hypothesis: There will be a greater improvement in overall FSFI with PTNS as compared to MT.

Secondary aims:

Aim 2: To determine if improvement in female sexual function with percutaneous tibial nerve stimulation or medical therapy is correlated with improvement in urinary symptoms as measured by the OAB-q questionnaire.

Hypothesis: Improvement in urinary symptoms will be correlated with improvement in sexual function but that the difference in FSFI between groups will not be solely attributable to differences in urinary symptom improvement.

Aim 3: To determine if changes in sexual function are greater with beta agonist medications as compared to anticholinergic medications.

Hypothesis: Beta agonists will result in improved sexual function as compared to anticholinergics.

Aim 4: To determine if those patients with female sexual dysfunction as defined as an overall FSFI score below 26.5 have greater improvements than those without.

Hypothesis: Patients with female sexual dysfunction will have a greater improvement in FSFI than those without.

Female sexual dysfunction (FSD) affects approximately 45% of women with an even greater incidence reported in women with overactive bladder symptoms, despite this there is a lack of FDA approved treatments for sexual dysfunction in this population. Female sexual function is complex and can be affected by pain, depression, and comorbidities as well as bowel and bladder function. There are numerous treatments for women with overactive bladder (OAB) defined as urinary urgency, frequency, urge urinary incontinence (UUI) and nocturia. These treatments include medical therapy (MT) with anticholinergics and beta agonists and neuromodulation via implantable sacral nerve stimulator (SNM) and percutaneous tibial nerve stimulation (PTNS). Sexual function, which can be measured by the Female Sexual Function Index (FSFI) has been shown to improve with both neuromodulation and anticholinergic therapy, although less is known about the effects of beta agonists. The purpose of this study is to examine the comparative effectiveness of neuromodulation via percutaneous tibial nerve stimulation and medical therapy with anticholinergics or beta-agonists in improving female sexual function. Additionally this study will assess whether improvement in sexual function is correlated with improvement in urinary symptoms. Furthermore the effectiveness of anticholinergics as compared to beta agonists with respect to changes in sexual function will be examined. Lastly patients with sexual dysfunction will be comapred to those without to determine if patients with female sexual dysfunction have greater improvements than those without, as this may open the door to future studies using PTNS for the primary indication of female sexual dysfunction. Enhanced understanding of the effects of neuromodulation and medical therapy on sexual function may allow for improved patient selection and better outcomes which may lead to widespread use of neuromodulation for female sexual dysfunction.

This is a prospective multi-center cohort study organized through the American Urogynecological Society Fellows Pelvic Research Network comparing changes in sexual function in women undergoing PTNS or MT for OAB/UUI. Recruitment is being conducted at MedStar Washington Hospital Center, MedStar Franklin Square, Indiana University, University of Texas Southwestern, University of Louisville and the University of Oklahoma. Potential subjects are adult women presenting to a urogynecology clinic for symptoms of overactive bladder such as urgency and UUI. Eligible subjects must report urinary urgency or urge incontinence and be recommended for treatment with medical therapy (with anticholinergic or beta agonist) or PTNS by the treating physician. Potential subjects are approached by their treating physician in the context of a private clinical visit regarding enrollment. Women who enroll are asked to complete the validated OAB-q, FSFI, Beck Depression Inventory and a visual analog pain scale prior to therapy and then again after twelve weeks of therapy. These forms may be completed in person on paper or via the online RedCap database. Demographic data including age, comorbidities and menopausal status are extracted from the medical record.

The primary endpoint of the study is improvement in overall FSFI score which is hypothesized to be greater in the PTNS group. Sample size calculations were conducted using http://clincalc.com/stats/samplesize.aspx with the primary endpoint of FSFI assessed as a continuous variable. Group sample sizes of 63 per group (total 126 patients) will be necessary to detect a clinically relevant difference of 5 points in FSFI assuming standard deviation of 10 and achieve a power of 80%, alpha=0.05. By incorporating a 10% loss to follow-up rate, the plan is to to recruit 70 patients per group, with a total of 140 patients. Because approximately 45% of patients with OAB will have FSD as determined by an FSFI score below 26.5, the study may include up to 312 patients in the study. A planned interim analysis will be conducted comparing patients receiving anticholinergics and those receiving beta agonists. This will be conducted once 63 patients receiving anticholinergics and 63 receiving beta agonists have completed the study. This will address Aim 3. A Mann-Whitney U test will be used to compare FSFI between patients receiving anticholinergics and beta agonists.

Data Collection and Transmission:

Potential subjects will be approached by their treating physician in the context of a private clinical visit regarding enrollment in the study. After discussion of the risks and benefits and obtaining written informed consent, each subject will be assigned a participant identification number (ID). Those patients who express interest but are unable to sign consent in the context of an office visit due to time constraints will be contacted via telephone to complete the consent process; once consent is obtained these patients will have the option of completing paper questionnaires which will be mailed to them or online questionnaires which they will receive through a secured email link. Treating physicians and investigators will monitor patients at clinic visits. Case report forms will be generated for each subject and completed by the investigator or study coordinator at each site, these will then be entered by the investigator or study coordinator into a password protected REDCap database with each patient identified only by ID. Patients will be asked to complete questionnaires in the setting of clinic visits to minimize mailings and their potential for privacy breach. Mailing of questionnaires will only be used if patients are unable to return to clinic for follow up; forms may also be returned via fax or secure email. Patients may also complete questionnaires online directly in the REDCap database. Patients will be encouraged to complete forms in REDCap to minimize the potential for transcription error and breach of privacy. For those patients who cannot mail the forms or access them online, they may be completed via phone with an investigator or study coordinator. Original case report forms and questionnaires will be securely maintained on site in a locked file cabinet within a locked office. MedStar Washington Hospital Center will be the Data Collecting Center (DCC). Copies of the case report forms and questionnaires will be forwarded by courier or fax to the DCC with participant ID number visible and personal information obscured. The following interim data will be monitored via review of the database at scheduled six-month intervals by the PI: accrual rate, patient adherence, adverse events and accuracy and completeness of the data.

ELIGIBILITY:
Inclusion Criteria:

* Female patients greater than 18 years of age
* Symptomatology of urinary urgency or urge incontinence planning to undergo MT or PTNS. Patients must meet a threshold bother defined by a positive response and bother of "somewhat, quite a bit, a great deal, or a very great deal" to questions #2, #3 or #8 on the OAB-q regarding urinary urgency and urgency incontinence.
* Patients may have tried other medication for overactive bladder in the past but should be off therapy for at least one month
* Patients must be currently sexually active with sexual activity within the past month and plans to continue for the duration of the study. Sexual activity, as defined in the FSFI questionnaire, may include caressing, foreplay, masturbation, and vaginal intercourse.

Exclusion Criteria:

* Contraindications to PTNS (skin, orthopedic or anatomical limitation that could prevent placement of PTNS electrode, presence of pacemaker)
* Contraindications to both anticholinergic and beta agonist therapy
* Current symptomatic UTI within past week
* Pregnant or planning to become pregnant
* Prior treatment with SNM, PTNS, onobotulinum toxin A or two medications (stopped for reasons unrelated to side effects)
* Diagnosed or suspected interstitial cystitis/painful bladder syndrome
* Diagnosis of neurogenic bladder
* Prolapse greater than Stage 2, pessary use or planned surgery for pelvic floor disorder during the study
* Planned simultaneous treatment with both PTNS and MT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Adult women presenting to a urology or urogynecology clinic for symptoms of overactive bladder such as urgency and UUI. Eligible subjects must report urinary urgency or urge incontinence and be recommended for treatment with medical therapy (with anticholinergic or beta agonist) or PTNS by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
overall FSFI | After 12 weeks
  Continuous variable

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gutman, MD, Principal Investigator — Medstar Health Research Institute
Locations (5):
- United States (5):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Oklahoma University, Oklahoma City, Oklahoma
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT03500146/Prot_SAP_001.pdf